CLINICAL TRIAL: NCT03336801
Title: The Effect of Propofol and Sevoflurane Anesthesia on Renal Function in Patients Undergoing Back Surgery
Brief Title: The Effect of Propofol or Sevoflurane on Renal Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Robert Frithiof, MD PhD, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ANIMAL-523-2014-2569
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Acute Kidney Injury; Anesthesia
Keywords: sevoflurane; propofol
MeSH Terms: conditions — Acute Kidney Injury | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: Patients are randomized into one of two treatment groups which during surgery receives one of two different anesthetic agents. The two groups are then compared to each other.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sevoflurane (Active Comparator): Intervention Back surgery and sevoflurane.
  Interventions: Procedure: Back Surgery; Drug: Sevoflurane
- Propofol (Active Comparator): Intervention Back surgery and propofol.
  Interventions: Procedure: Back Surgery; Drug: Propofol

INTERVENTIONS:
Procedure: Back Surgery — All patients undergo basic back surgery.
Drug: Propofol — Anesthesia on propofol alone.
  Arms: Propofol
Drug: Sevoflurane — Anesthesia on sevoflurane alone.
  Arms: Sevoflurane

SUMMARY:
This study investigates the role of the anesthetic agents propofol and sevoflurane on renal function in otherwise healthy patients undergoing basic back surgery.

DETAILED DESCRIPTION:
Water-sodium homeostasis is central for anyone undergoing surgery, and can therefore affect surgical outcome, level of postoperative care and the length of hospital stay. Too much or too little fluid during surgery can affect the patients negatively. The kidneys play an imperative role in the regulation of water and sodium homeostasis, however there are lack of knowledge in how the anesthesia per se affects renal function. Previous studies have shown that volatile anesthetic agents such as sevoflurane can cause fluid retention. Why this happens is not completely known.

We are now investigating the different affects of sevoflurane and propofol anesthesia on renal function in patients undergoing basic back surgery to elucidate if there is a difference in the risk of developing acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled back surgery

Exclusion Criteria:

* American Association of Anesthesiology class 1-3
* American Heart Association class >3
* BMI >37
* Insulin treated diabetes
* Pregnancy or breast feeding
* Sensistivity/allergy against anesthetic agents
* Inadequate understanding about the study
* Depressed kidney function and/or AKI
* Depressed liver function
* Genetic malignant hyperthermia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Change in urine output | 24 hours
  Urine output (ml/min) changes during anesthesia, in postoperative care and in the ward unit. Changes will be assessed with AKIN RIFLE and by comparison between the different groups.
Change in serum creatinine levels | 24 hours
  Changes in serum creatinine levels during anesthesia, in postoperative care and in the ward unit. Changes will be assessed with AKIN RIFLE and by comparison between the different groups.
Change in creatinine clearance | 24 hours
  Creatinine clearance changes during anesthesia, in postoperative care and in the ward unit. Changes will be assessed with AKIN RIFLE and by comparison between the different groups.

SECONDARY OUTCOMES:
Changes in electrolytes | 24 hours
  Changes in serum and urinary electrolytes (sodium and potassium) will be measured during anesthesia, in postoperative care and in the ward unit.
Changes in hormone levels | 24 hours
  The hormones angiotensin II, anti diuretic hormone and aldosterone will be measured during anesthesia, in postoperative care and in the ward unit.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Franzén, PhD, Principal Investigator — Uppsala University, Department of Anesthesiology and Intensive Care; Robert Frithiof, MD PhD, Study Director — Uppsala University, Department of Anesthesiology and Intensive Care
Locations (1):
- Akademiska sjukhuset, Centraloperation, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No